CLINICAL TRIAL: NCT05619874
Title: Effects of Two Virtual High-intensity Functional Circuit Training Programs on Intra-abdominal Fat, Body Composition, Health-related Quality of Life, and Some Components of Physical Fitness in Adults With Abdominal Obesity
Brief Title: Effects of Two Virtual HIFCT Programs in Adults With Abdominal Obesity
Acronym: HIFCT-V
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended due to the inability to complete the sample after more than a year of attempts. Various adherence strategies were tested, but adherence to the interventions remained too low.
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victor Hugo Arboleda Serna, Principal Investigator, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Virtual HIFCT-UdeA-SENA_DC
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: High-intensity functional circuit training; Virtual exercise; Obesity; Intra-abdominal fat; Waist circumference; Body composition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFCT-S (Experimental): For sessions 7 to 14, a concentrated circuit divided into four blocks of three exercises will be carried out, with a duration of 40 seconds per exercise with no rest between them. A rest of 120 seconds will be given at the end of each block, and a rest of the same time at the end of the first set. Two sets will be executed, which will result in a total time of 30 minutes including rest. For sessions 15 to 30, four blocks of two exercises will be performed, with a duration of 60 seconds per exercise, with no rest between them. The rest between blocks will be 120 seconds. Two sets will be performed, for a total time of 30 minutes including breaks. The exercises will be performed at speeds between 35 and 75 bpm. The intensity will be between 80% - 90% (8-9 RPE).
  Interventions: Behavioral: HIFCT-S
- HIFCT-P (Active Comparator): For sessions 7 to 14, a concentrated circuit divided into two blocks of six exercises will be carried out, with a duration of 60 seconds per exercise with no rest between them. A rest of 120 seconds will be given at the end of each block, and a rest of the same time at the end of the first set. Two sets will be executed, which will result in a total time of 30 minutes including rest.
  For sessions 15 to 30, five blocks of two exercises will be performed, with a duration of 120 seconds per exercise, with no rest between them. The rest between blocks will be 120 seconds. The total time per block is four minutes, for a total time of 30 minutes including breaks. The exercises will be performed at speeds between 35 and 75 bpm. The intensity will be between 80% - 90% (8-9 RPE).
  Interventions: Behavioral: HIFCT-P

INTERVENTIONS:
Behavioral: HIFCT-S — A functional circuit training of 30 sessions will be carried out as follows:
  * Sessions 1 to 6: General circuit (two series) composed of four blocks of three exercises.
  * Sessions 7 to 14: Concentrated circuit (two sets) composed of four blocks of three exercises of greater complexity than the exercises of the general circuit.
  * Sessions 15 to 22: Circuit by blocks (two sets) composed of four blocks of two exercises of greater complexity than the exercises from sessions 7 to 14.
  * Sessions 23 to 30: Circuit by blocks (two sets) composed of four blocks of two exercises of greater complexity than the exercises from sessions 15 to 22.
  Arms: HIFCT-S
Behavioral: HIFCT-P — A functional circuit training of 30 sessions will be carried out as follows:
  * Sessions 1 to 6: General circuit (two series) composed of two blocks of 6 exercises.
  * Sessions 7 to 14: Concentrated circuit (two sets) composed of two blocks of 6 exercises of greater complexity than the exercises of the general circuit.
  * Sessions 15 to 22: Circuit by blocks (single set) composed of five blocks of two exercises of greater complexity than the exercises from sessions 7 to 14.
  * Sessions 23 to 30: Circuit by blocks (single set) composed of five blocks of two exercises of greater complexity than the exercises from sessions 15 to 22.
  Arms: HIFCT-P

SUMMARY:
It is estimated that by 2030 one in five women and one in seven men will be obese, equivalent to more than 1 billion people around the world. It should be noted that the largest number of people with obesity live in countries with low and moderate-income. In 2019, more than 160 million years of healthy life were lost in the world, due to a high body mass index (BMI), this represents more than 20% of all years of healthy life lost due to chronic diseases. Therefore, it is essential to stop the increase in obesity and reduce it at all ages, which demands comprehensive actions at the global level. Scientific evidence suggests that people with a normal BMI, but with abdominal obesity, have a higher mortality risk compared to those with a similar or even higher BMI. In addition, visceral adiposity has been associated with worse survival and with colorectal cancer.

Several methods of physical exercise have been used to counteract the adverse effects of obesity, including high-intensity functional circuit training (HIFCT). Scientific evidence indicates that HIFCT reduces fat mass, body mass, BMI, and waist circumference and improves muscle strength, maximal oxygen uptake, and health-related quality of life in overweight, obese, inactive, and with other diseases. However, no research assessed intra-abdominal fat (IAF), which, more than subcutaneous fat, is associated with cardiovascular risk factors. In addition, these studies had important methodological limitations. Therefore, the primary purpose of this study is to identify the effect of two HIFCT protocols, prolonged load (HIFCT-P) and short load (HIFCT-S), performed in a virtual environment for ten weeks on intra-abdominal fat in people between 18-40 years-old with abdominal obesity.

DETAILED DESCRIPTION:
A randomized controlled trial with parallel arms (HIFCT-P and HIFCT-C) based on a non-inferiority hypothesis comparing two proportions. Each participant will carry out 30 sessions, three times a week, in a virtual environment. General, concentrated, and block circuits will be used, with the same exercises, but with different load distribution and different order between them. Both HIFCT-P and HIFCT-S will carry out six initial adaptation sessions through a general circuit composed of 12 exercises. Different muscle groups will be alternated. The exercises will be performed at speeds between 35 and 55 beats per minute (bpm), to ensure intensities between 50% - 60% in sessions 1 to 3, and between 70% - 80% in sessions 4 to 6. The Modified Borg Rating of Perceived Exertion Scale (RPE) will be used to control intensities. From session seven to session 30, HIFCT-P and HIFCT-S will perform the same exercises but with a different load distribution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men.
* Physical activity (<600 to ≤1500 MET/min/wk).
* Waist circumference (≥87cm).

Exclusion Criteria:

* Have performed high intensity exercises or HIFCT in the last two months.
* Smoking.
* History of cardiovascular disease.
* History of coronary heart disease.
* Pregnancy.
* Breast-feeding women.
* Psychological, neuromotor, and/or osteo-muscular conditions that may affect participation in an exercise program.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Change in intra-abdominal fat | Baseline and 10-weeks
  Body Composition Analyzer Seca mBCA 515. The measurement results allow estimating intra-abdominal fat in liters. Values <27 L are considered normal, >27 L to <43 L are considered elevated, and ≥43 L are considered high. Individuals will be instructed to wear light clothing, and stand barefoot on the device, following manufacturer protocols.All assessments will take place at the same time of day.

SECONDARY OUTCOMES:
Change in waist circumference | Baseline and 10-weeks
  A flexible tape measure: Waist circumference will be measured following standard procedures, at the mid-point between the lower costal edge and the iliac crest. (Klein et al., 2007 https://doi.org/10.1093/ajcn/85.5.1197)

OTHER OUTCOMES:
Fat mass, fat-free mass, whole-body and segmental skeletal muscle mass. | Baseline and 10-weeks
  Body Composition Analyzer Seca mBCA 515. Individuals will be instructed to wear light clothing, and stand barefoot on the device, following manufacturer protocols. All assessments will take place at the same time of day.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Formación en Actividad Física y Cultura-SENA Distrito Capital, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No